CLINICAL TRIAL: NCT06231004
Title: A Study on the Correlation Between the Microbiome and Type 2 Inflammatory Diseases of Chronic Rhinosinusitis With Nasal Polyps (CRSwNP)
Brief Title: Correlation Between the Microbiome and Type 2 Inflammatory Diseases of CRSwNP
Status: Not yet recruiting | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Cheng Lei, Professor， PhD, The First Affiliated Hospital with Nanjing Medical University
Other Study IDs: Microbiome and CRSwNP
Record Dates: First submitted 2024-01-21; First posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Chronic Rhinosinusitis With Nasal Polyps (CRSwNP)
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Collection of feces, saliva, plasma, nasal microorganisms， tonsil microorganisms, nasal exfoliated cells and nasal secretions
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental group: Take glucocorticosteroid at once in the morning and use the following course of treatment: 6 tablets/day for 7 days-- 5 tablets/day for 2 days-- 4 tablets/day for 2 days-- 3 tablets/day for 2 days-- 2 tablets/day for 2 days-- 1 tablets/day for 2 days--surgery
  Interventions: Procedure: glucocorticosteroid and surgery

INTERVENTIONS:
Procedure: glucocorticosteroid and surgery — Take glucocorticosteroid at once in the morning and use the following course of treatment: 6 tablets/day for 7 days-- 5 tablets/day for 2 days-- 4 tablets/day for 2 days-- 3 tablets/day for 2 days-- 2 tablets/day for 2 days-- 1 tablets/day for 2 days--surgery

SUMMARY:
Nasal microorganisms, exfoliated cells, nasal secretions, fetal microorganisms and blood were collected from patients with chronic sinusitis with nasal polyps before medication. Nasal polyp tissues of the patients were clamped for pathologic biopsy in the outpatient clinic. Methylprednisolone was then administered to the patients for 17 days, and the nasal microbial changes were observed after the administration of the drug. Patients underwent surgical treatment after the administration of the drug, and postoperative patients were followed up for a long period of time until polyp recurrence. During the follow-up, the microorganisms in the patients' postoperative nasal cavities were collected and the postoperative microbial changes were recorded

DETAILED DESCRIPTION:
In this study, we retrospectively collected pathologic paraffin specimens and patient information from previous cases of sinusitis with nasal polyps, and prospectively collected specimens from newly enrolled patients with nasal polyps.

ELIGIBILITY:
Inclusion Criteria:

- The diagnosis of CRSwNP was based on EPOS20201 ECRSwNP was defined as EO accounting for more than 27% of the total infiltration Subjects undergoing septoplasty due to anatomical variations served as controls Discontinuation of steroid (oral or aerosol) and antileukotriene therapy for at least 4 weeks prior to biopsy or surgery

Exclusion Criteria:

- Exclude patients with a diagnosis of posterior maxillary sinus polyps, cystic fibrosis, allergic fungal sinusitis, primary ciliary dyskinesia, allergic rhinitis, immune deficiency, or coagulopathy Exclusion of patients with aspirin intolerance (AERD) Exclude smokers Exclude pregnant women

Healthy Volunteers:

Only patients with deviated septum without any other nasal diseases served as a control group, and the participants in this group were not treated with corticosteroids and went in for septal correction. The rest of the criteria were the same

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All Patients in the First Affiliated Hospital, Nanjing Medical University and volunteering for this study
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-01-22 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2032-09-01 (Estimated)

PRIMARY OUTCOMES:
Nasal polyp size after glucocorticosteroid | 17days
  Patients who did not have a reduction of more than 1 polyp score based on the NPSS system after glucocorticoid therapy were defined as glucocorticoid nonresponders
endoscopic evidence of returned polyposis | 3 years
  endoscopic evidence of returned polyposis, together with 1 or more bothersome symptoms (nasal obstruction, rhinorrhea, headache/facial pain, smell abnormalities, and sleep disturbance/fatigue) lasting at least 1 week even after receiving appropriate intranasal GC treatment

CONTACTS AND LOCATIONS:
Overall Officials: Lei Cheng, Study Director — The First Affiliated Hospital, Nanjing Medical University

IPD SHARING:
Plan to Share IPD: No
All the individual participant data only available to reasearchers participated in this study